CLINICAL TRIAL: NCT02971514
Title: Comparative Efficacy of Dental Flossing Before or After Tooth Brushing on Interproximal Plaque Reduction and Fluoride Retention in That Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fatemeh Mazhari, Associate professor od Pedodontics, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 920200
Record Dates: First submitted 2016-11-11; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Floss-Brush group (Experimental): The participants flossed first followed by brushing
  Interventions: Behavioral: Flossing before Brushing
- Brush-Floss group (Active Comparator): They used dental floss after brushing
  Interventions: Behavioral: Brushing before Flossing

INTERVENTIONS:
Behavioral: Flossing before Brushing
  Arms: Floss-Brush group
Behavioral: Brushing before Flossing
  Arms: Brush-Floss group

SUMMARY:
This randomized controlled crossover trial conducted on 25 dental students. in the preliminary session each volunteer was given a toothbrush(Trisa, soft, Switzerland) and toothpaste(Pooneh, Iran) and Dental Floss( Mina, Iran)to use during the study, and they were instructed the proper techniques of brushing and flossing.The study was performed in two treatment sessions and a 48 hour washout period. They passed through the sessions in a randomized sequence. After prophylaxis with rubber cup, they were asked to discontinue all oral hygiene for 24 hour. At the first session , they flossed first followed by brushing (floss-brush group) and at the other session they used dental floss after brushing (brush-floss group) . At each session, before and after brushing and flossing , Dental plaque reduction was assessed using Rustogi Modified Navi Plaque Index. Interdental plaque was collected for measuring fluoride. Differences between the two groups were analyzed with mixed model test.

ELIGIBILITY:
Inclusion Criteria:

* Dental students with 16 teeth in each jaw who had Normal salivary volume No active caries No medicine which could be affect salivary secretion No fluoride consumption in the last two weeks No Antibiotic consumption in the last 4 weeks

Exclusion Criteria:

* Any systemic diseases Periodontal diseases Crowding

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Dental plaque reduction | immediately Before brushing/ flossing and immediately after these procedures
  Dental plaque assessed using a scale known as: "Rustogi Modified Navy Plaque Index"

SECONDARY OUTCOMES:
fluoride concentration in Interdental plaque | Immediately after toothbrushing /flossing interdental plaque was collected for fluoride measurement
  fluoride concentration measured using ppm scale (microgram/milliliter)

CONTACTS AND LOCATIONS:
Locations (1):
- Amir Moeintaghavi, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- [Derived] Mazhari F, Boskabady M, Moeintaghavi A, Habibi A. The effect of toothbrushing and flossing sequence on interdental plaque reduction and fluoride retention: A randomized controlled clinical trial. J Periodontol. 2018 Jul;89(7):824-832. doi: 10.1002/JPER.17-0149. Epub 2018 Jul 20. PMID 29741239